CLINICAL TRIAL: NCT00524498
Title: A Phase II Study of a Continuous Hepatic Arterial Infusion Combination Therapy With OPC-18 and 5-FU in Patients With Highly Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 018-06-002
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: OPC-18; Interferon-alpha; Fluorouracil
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): FAIT
  Interventions: Drug: OPC-18
- B (Active Comparator): BST
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: OPC-18 — OPC-18: 500IU * 3 times a week, sc 5-FU : 500mg infusion for 5days into hepatic artery
  Arms: A
Drug: cisplatin — infusion into hepatic artery with cisplatin 10mg and 5-FU 250mg a day
  Other Names: low-dose FP treatment
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a continuous hepatic arterial infusion combination therapy with OPC-18 and 5-FU versus BST in patients with highly advanced hepatocellular carcinoma for which resection therapy or local therapy is inapplicable due to advanced vascular invasion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are histologically or clinically (diagnostic imaging and tumor marker) diagnosed with hepatocellular carcinoma
* Patients with a measurable lesion by contrast CT
* Patients with no remote metastasis (extrahepatic metastasis), confirmed by X-ray, CT, MRI, or other means if necessary
* Patients who have not previously received intra-arterial hepatic chemotherapy

Exclusion Criteria:

* Patients receiving the herbal medicine shosaikoto
* Patients with autoimmune hepatitis
* Patients with a history of hypersensitivity to OPC-18 or other interferon preparations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Antitumor effect (tumor size reduction) | every 4 weeks

SECONDARY OUTCOMES:
Disease control rate Overall survival Progression-free survival | every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Divsion of New Product Development
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region